CLINICAL TRIAL: NCT06534060
Title: A Phase 2, Open-label, Multicenter Study of MB-105 in Patients With CD5 Positive (CD5+) Relapsed / Refractory T-cell Lymphoma (r/r TCL).
Brief Title: MB-105 in Patients With CD5 Positive T-cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: March Biosciences Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MB-105-201
Record Dates: First submitted 2024-07-25; First posted 2024-08-02 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Lymphoma, T-Cell
Keywords: MB-105-201
MeSH Terms: conditions — Lymphoma, T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Other): This is a single arm, two-stage, Phase 2, open-label, multicenter study.
  Interventions: Biological: Genetic: MB-105

INTERVENTIONS:
Biological: Genetic: MB-105 — MB-105 is a CAR T-cell therapy that consists of autologous T-cells that express a CD5 CAR.

SUMMARY:
This is a single arm, two-stage, Phase 2, open-label, multicenter study of MB-105 in patients with CD5 Positive (CD5+) Relapsed / Refractory T-cell Lymphoma (r/r TCL). This study will apply a Simon two-stage optimal design.

DETAILED DESCRIPTION:
The first stage of the Simon two-stage design will enroll approximately 15 evaluable patients. Once the first 6 patients are enrolled, have received one dose of MB-105 at the recommended phase 2 dose (RP2D), and completed at least up to Day 30 of the study, the Independent Data Monitoring Committee (IDMC) will perform a safety analysis. The IDMC will use this analysis to confirm that the RP2D selected for this Phase 2 study is the appropriate dose of MB-105 for further clinical evaluation. The IDMC will either recommend continuing the remainder of the study at the fixed dose of 50 million (5 x 107) Chimeric antigen receptor (CAR) positive cells or recommend other actions, which could include repeating the safety run-in with either a lower or higher dose. The IDMC will not recommend a MB-105 dose greater than those found safe in the phase 1 study. During the safety analysis period after the 6th patient is treated and awaiting data analysis, patients will continue to be screened but not dosed until the IDMC recommendation is made.

If the IDMC confirms the suggested RP2D is the appropriate dose for further clinical evaluation, the study will enroll an additional 9 patients to complete 15 total patients for Stage 1 to obtain a preliminary estimate of response rate per Lugano criteria for peripheral T-cell lymphoma (PTCL) and 2022 Global criteria for cutaneous cases (CTCL). At the end of Stage 1, defined as when the last patient enrolled completes study visits up to Day 56, including efficacy assessment, the IDMC will convene to review all available Stage 1 data and recommend continuation to Stage 2 or closure of enrollment.

Stage 2 will enroll approximately 31 patients, for a total of 46 patients in the study. During Stage 2 the IDMC will convene at least once every 6 months to review safety and efficacy on an ongoing basis. No formal interim analysis is planned after the end of Stage 1, but since this is an open-label study, interim data extracts may be performed to support abstract submissions, presentations, or regulatory discussions. The study will end once the last patient completes at least 12 months of follow-up and end of study (EOS) visit. After EOS, all patients will be asked to participate in a separate long term follow-up (LTFU) study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age.
2. Patients with r/r TCL per WHO 2022 criteria.

   1. r/r CTCL that has failed ≥ 2 prior lines of standard of care (SoC) therapy.
   2. r/r PTCL that has failed ≥ 1 prior lines of SoC therapy. Note: patients with CD30+ disease should have received brentuximab vedotin.
3. Has available tumor tissue or is willing to undergo a biopsy procedure.
4. CD5 positivity confirmed by local laboratory using an approved diagnostic test or LDT. CD5 positivity is currently defined as having ≥ 50% CD5 expression. An exploratory cohort will enroll patients with CD5 expression below 50%.
5. Karnofsky performance score ≥ 70% or higher.
6. Prior CAR T-cell therapy must have occurred > 60 days prior to study enrollment and must have no evidence of CAR persistence.
7. Measurable or detectable disease

   1. PTCL per Lugano criteria
   2. CTCL per Global (ISCL/EORTC/USCCL) criteria.
8. Prior autologous or allogenic hematopoietic stem cell transplant (HSCT) must have occurred more than 60 days prior to study enrollment.
9. Adequate bone marrow function defined as:

   1. Absolute neutrophil count (ANC) ≥ 1500/μL (≥ 1000/μL for patients with prior HSCT or marrow involvement)
   2. Absolute lymphocyte count ≥200 cells/μL
   3. Hemoglobin ≥ 8 g/dL (transfusion permitted)
   4. Platelet count ≥ 75 000/μL (≥50 000/μL for patients with marrow involvement).
10. Organ function as follows:

    1. Cardiac: left ventricular ejection fraction (LVEF) ≥ 50% by Echo or radionuclide scan.
    2. Pulmonary: oxygen saturation ≥ 92% (room air).
    3. Renal: calculated creatinine clearance > 30 mL/min.
    4. Liver:

       * Total bilirubin < 1.5 x ULN (< 2 × upper limit of normal (ULN)) if liver involvement).
       * If no liver involvement and total bilirubin ≥1.5 x ≤ ULN, direct bilirubin < ULN (Gilbert syndrome)
       * Aspartate aminotransferase / alanine aminotransferase < 3 × ULN (5 x ULN if liver involvement).
       * Albumin > 2.5 g/dL.
11. For females of childbearing potential (defined as < 24 months of amenorrhea or not surgically sterile [absence of ovaries and/or uterus]), a negative serum pregnancy test must be documented at screening, and prior to lymphodepletion (conditioning).
12. For females of childbearing potential and males, a highly effective method of contraception together with a barrier method must be used from the start of lymphodepletion (conditioning) and for at least 12 months after the last dose of study agent.

Exclusion Criteria:

1. Sezary syndrome. For other tumor types, if there is a suspicion of significant circulating disease at time of leukapheresis, discuss eligibility with medical monitor prior to proceeding.
2. Contraindication to leukapheresis.
3. Prior treatment with any CD5-targeted therapy.
4. Any evidence of the following active viral infections:

   1. HIV infection.
   2. Chronic hepatitis B virus (cHBV) infection with detectable viral load. Patients with cHBV, who are receiving anti-viral prophylaxis, may be enrolled if they are asymptomatic for >5 days prior to signing informed consent (ICF).
   3. Hepatitis C (HCV) infection with detectable viral load. Patients cured of HCV may be enrolled.
5. Presence of any active, uncontrolled systemic bacterial, viral or fungal infection requiring intravenous (IV) anti-infectives, including clinically significant viral infection or uncontrolled viral reactivation of Epstein-Barr virus, Cytomegalovirus, Adenovirus, BK-virus, or Human herpesvirus 6. If treated with anti-infective agents, patients must be asymptomatic for >5 days prior to enrollment.
6. History of any malignancy within 2 years with the exception of cured stage 1 cancers or CIS and potentially indolent cancers not requiring active treatment or controlled with hormone therapy. Discuss patients with indolent cancers with the medical monitor.
7. History of hypersensitivity reactions to products containing murine proteins.
8. Active CNS lymphoma.
9. Evidence of acute graft versus host disease (aGVHD) > Grade 2 Mount Sinai Acute GVHD International Consortium (MAGIC) or chronic GVHD > mild (NIH) requiring ongoing systemic steroids and/or multiagent therapy.
10. Patients who have received systemic immunosuppressive therapy for treatment of GVHD within 28 days of leukapheresis.
11. Currently requiring systemic corticosteroid therapy (10 mg/day or less of prednisone or equivalent doses of other systemic steroids are allowed for control of non-exclusionary pre-existing conditions). A 2-week washout is required prior to leukapheresis and prior to lymphodepletion for patients on > 10 mg/day prednisone equivalent.
12. Patients who have received donor lymphocyte infusions within 28 days of MB-105 infusion.
13. Comorbidity that would impair the patient's ability to receive or tolerate MB-105 and/or affect participation in the study:

    1. History of cardio- or cerebrovascular disease including myocardial infarction, unstable angina, or congestive heart failure (NYHA class III-IV) within 6 months or cerebrovascular accident (CVA; stroke) within 12 months prior to informed consent.
    2. History of central nervous system (CNS) disorder(s) such as an uncontrolled seizure disorder, dementia, cerebellar disease, or any autoimmune disease with CNS involvement.
    3. Any serious underlying medical or psychiatric condition deemed by the investigator and medical monitor to be exclusionary due to risk to the patient or to protocol compliance.
14. History of autoimmune disorders, including rheumatic diseases and thyroid disorders (though patients with a history of thyroid disease who have undergone successful therapy may be suitable). Exemptions for mild or limited disease may be granted after discussion between the Investigator and sponsor's medical monitor.
15. Participated in active treatment on other interventional research clinical trials < 30 days before enrollment (participation in follow-up permitted). Contact the medical monitor to discuss prior experimental agents targeting the T cell lineage and the appropriate washout period.
16. Received bendamustine prior to enrollment (unless received an allo-HSCT in the interim).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | 26 months
  Incidence, severity, causal relationship of AEs
Objective response rate (ORR) | 26 months
  Best objective response rate (ORR) per independent central review as defined by rate of complete response (CR) and PR using the 2014 Lugano criteria and 2022 Global criteria.

SECONDARY OUTCOMES:
Duration of response (DOR) | 26 months
  Duration of Response (DOR), defined as time from first observation of response to the time of disease progression or death, whichever comes first (per investigator and by central review).
Progression-free survival (PFS) | 26 months
  Progression-free survival (PFS), defined as time from administration of MB-105 to the time of disease progression or death, whichever comes first (per investigator and by central review).
Incidence of adverse events during the safety monitoring period for acute toxicities | 26 months
  * All AEs from leukapheresis up to Day 30.
  * Related AEs from MB-105 infusion to Day 90 (i.e. excluding only AEs that are clearly an expected event from underlying condition or non-study related treatment).
  * SAEs and all-cause mortality from MB-105 infusion to EOS at Month 24.
Overall survival (OS) | 26 months
  Overall survival (OS), defined as time from administration of MB-105 to death.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Bexon, MD, CMO, Study Chair — March Bio
Locations (12):
- United States (12):
  - University of San Diego (UCSD)-Moores Cancer Center, San Diego, California
  - SCRI - Colorado Blood Cancer Institute (CBCI), Denver, Colorado
  - Moffitt Cancer Center Magnolia Campus, Tampa, Florida
  - University of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Nebraska, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregan Health & Science University, Portland, Oregon
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas